CLINICAL TRIAL: NCT03862235
Title: Decreased Myocardial Native T1 Times and Impaired Myocardial Contractility in Young Anabolic Androgenic Steroids Users
Brief Title: Decreased T1 Times and Impaired Myocardial Contractility in Anabolic Androgenic Steroids Users
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Maria Janieire de Nazaré Nunes Alves, Principal Investigator, MD, PhD, University of Sao Paulo General Hospital
Other Study IDs: CMR- AnabolicSteroids
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Focal Fibrosis
Keywords: anabolic steroid; T1-mapping; cardiac structure
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anabolic androgenic steroids users: This group had been involved in strength training for at least 2 years, self-administering anabolic androgenic steroids in periodic cycles lasting from 8 to 12 weeks for at least 2 years with 2-4 cycles per year. All participants were on a cycle over the course of the study.
  Cardiovascular magnetic resonance (CMR) with late-gadolinium enhancement (LGE), cardiac T1-mapping and extracellular volume (ECV). Cardiac contractility was evaluated as cardiac strain by CMR (feature tracking) and transthoracic echocardiography (speckle tracking).
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance; Diagnostic Test: Transthoracic echocardiography
- Anabolic androgenic steroids nonusers: This group had been involved in strength training for at least 2 years and they have never took anabolic androgenic steroids.
  Cardiovascular magnetic resonance (CMR) with late-gadolinium enhancement (LGE), cardiac T1-mapping and extracellular volume (ECV). Cardiac contractility was evaluated as cardiac strain by CMR (feature tracking) and transthoracic echocardiography (speckle tracking).
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance; Diagnostic Test: Transthoracic echocardiography
- Sedentary control: This group were sedentary men without cardiovascular disease.
  Cardiovascular magnetic resonance (CMR) with late-gadolinium enhancement (LGE), cardiac T1-mapping and extracellular volume (ECV). Cardiac contractility was evaluated as cardiac strain by CMR (feature tracking) and transthoracic echocardiography (speckle tracking).
  Interventions: Diagnostic Test: Cardiovascular Magnetic Resonance; Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Cardiovascular Magnetic Resonance — The patients underwent to CMR examination on a Philips Achieve 1.5 device. Images were acquired coupled to the electrocardiogram and during respiratory pause, in four chambers, short axis and long axis of the left ventricle, in the same exact location in different sequences. A gradient - echo sequence (steady-state free precession) was used to evaluate cardiac function (functional evaluation). We will also evaluate T1 weighted images (T1 -relaxation times) and T2, performed sequentially, through spin-echo pulse (black-blood), triple inversion recovery sequence, for the morphological evaluation
Diagnostic Test: Transthoracic echocardiography — The images were collected by the Vivid E9. The patients were submitted to one-dimensional (M-mode), two-dimensional (B-mode), and three-dimensional (three-dimensional) echocardiographic studies. The images obtained were associated with pulsed, continuous and color Doppler.

SUMMARY:
Anabolic androgenic steroids (AAS) abuse may have a toxic on myocardium that could lead to cardiac alterations. Clinical cases reported myocardial fibrosis in AAS users. However, recent studies did not find myocardial fibrosis in AAS users using T1-mapping technique. The aim of this study was to evaluate cardiac structure by cardiovascular magnetic resonance (CMR) with late-gadolinium enhancement (LGE), cardiac T1-mapping and extracellular volume (ECV). We also evaluated the cardiac contractility in AAS users.

DETAILED DESCRIPTION:
Twenty strength-trained AAS users (AASU) age 29±5 yr, 20 age-matched strength-trained AAS nonusers (AASNU), and 10 sedentary controls (SC) were enrolled.

Cardiac structure was assessed by LGE, T1-mapping and ECV. Cardiac contractility was evaluated as cardiac strain by CMR (feature tracking) and echocardiography (speckle tracking)

ELIGIBILITY:
Inclusion Criteria:

* Anabolic androgenic steroids users and Anabolic androgenic steroids nonusers groups had been involved in strength training for at least 2 years;
* Anabolic androgenic steroids users should be self-administering anabolic androgenic steroids in periodic cycles lasting from 8 to 12 weeks for at least 2 years with 2-4 cycles per year;
* All anabolic androgenic steroids users were on a cycle over the course of the study;
* Sedentary control group: sedentary men without cardiovascular disease.

Exclusion Criteria:

* Smoking;
* Alcohol consumption;
* Use of diuretics and/or antihypertensive medications;
* Liver and kidney disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Anabolic androgenic steroids users and nonusers were recreational weightlifters or amateur bodybuilding athletes who were recruited from gymnasiums.
  Sedentary control group was recruited from community sample.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Cardiac T1-mapping | 1 day
  For the identification of microscopic interstitial fibrosis and the calculation of extracellular space volume (ECV) were use the T1-mapping technique, which use the Modified Lock-Locker (MOLLI) pulse sequence. It was performed for image acquisition, before contrast injection with 3 short-axis cuts, in order to define the baseline T1 of myocardium. The evaluation of the MOLLI sequence images at 4 different times has the objective of evaluating the recovery of T1 times after contrast injection, which allows, associated with hematocrit, the calculation of myocardial extracellular space that is directly related to fibrosis in validation studies with endomyocardial biopsy.

SECONDARY OUTCOMES:
Myocardial Contractility | 1 day
  To calculate the left ventricular function, the strain values were used. Using the speckle-tracking technique, the value of the global longitudinal strain (GLS) was extracted through the three apical views, later the mean of 17 myocardial segments was calculated. Normal value for GLS was set to -18%, although in the literature there is no standardized value. Circumferential and radial strain values were estimated by short-axis parasternal views.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Janieire NN Alves, MD, Principal Investigator — Heart Institute (InCor), University of Sao Paulo Medical School
Locations (1):
- Instituto do Coração do Hospital da Clínicas da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No